CLINICAL TRIAL: NCT00841243
Title: The Effects of Preventive Versus on Demand Nutritional Advice and Support on the Nutritional Status of Patients During Antiviral Therapy for Hepatitis C A Randomized, Multi Center Trial
Brief Title: Nutritional Support During Antiviral Therapy for Hepatitis C
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Dr K.J. van Erpecum, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-70
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Hepatitis C; Weight Loss
Keywords: Hepatitis C; Antiviral therapy; weight loss; dietary support; dietary advise
MeSH Terms: conditions — Hepatitis C; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nutritional advise/support (Active Comparator): Nutritional advise and support
  Interventions: Dietary Supplement: Nutrison (Nutricia)
- control (No Intervention): Control

INTERVENTIONS:
Dietary Supplement: Nutrison (Nutricia) — During 48 weeks of treatment, the patient will receive at T=0, 2, 4, 8, 12, 18, 24, 36, 48 weeks dietary advise combined with daily nutritional support in the form of a nutritional supplement drink at bedtime.
  Other Names: Nutridrink protein (Nutricia, The Netherlands)
  Arms: nutritional advise/support

SUMMARY:
Standard antiviral treatment consists of weekly injections with Peginterferon-α in combination with ribavirin. This treatment may lead to significant weight loss (7% within 24 weeks on average), with decreased quality of life. In this study the investigators will examine in 50 patients whether nutritional advise and support can prevent weight loss during antiviral therapy.

DETAILED DESCRIPTION:
Standard antiviral treatment consists of weekly injections with Peginterferon-α in combination with ribavirin. This therapy, however, leads to weight loss of approximately 7% in the first 24 weeks of therapy possibly related to impaired postprandial gastric emptying. Such rapid weight loss is a marker of deterioration of the nutritional status with increased risk of complications and reduced immunological barrier function. Deterioration of the nutritional status also exacerbates side effects of the antiviral treatment like fatigue and depression. As a result, the quality of life of these patients may decrease. In the current controlled, prospective, multicenter, study we primarily aim to compare the effects of preventative versus on demand nutritional advice in combination with nutritional support on reduction of weight loss in patients receiving standard antiviral therapy with PEG-interferon in combination with ribavirin. We will randomize patients for the preventative intervention with dietary consultation combined with dietary supplementation of a daily snack or the on demand dietary support group (only dietary follow up, no dietary advice or snack, standard care). In the on demand group, patients will be referred to the dietitian in case of weight loss of ≥ 5% or a BMI < 20 during antiviral therapy. Assuming that 60% reduction of weight loss during the first 24 weeks of treatment is clinically relevant, 2 x 25 patients need to be included (α=0.05, β=0.2: power=0.8 and a drop-out rate of 15%). Primary aim is to assess whether the intervention can decrease the amount of weight loss during therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hepatitis C
* Indication for antiviral therapy
* Age > 18 years
* Good understanding of Dutch or English language
* Informed consent

Exclusion Criteria:

* Co-infection with hepatitis B and/or HIV
* Significant non hepatic diseases
* Significant previous surgery of the gastro-intestinal tract
* Hepatocellular carcinoma or other current malignant disease
* BMI < 20

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Karel van Erpecum, Dr, Principal Investigator — UMC Utrecht
Locations (1):
- UMC, Utrecht, Netherlands

REFERENCES:
- [Background] Kruizenga HM, Wierdsma NJ, van Bokhorst MA, de van der Schueren, Haollander HJ, Jonkers-Schuitema CF, van der Heijden E, Melis GC, van Staveren WA. Screening of nutritional status in The Netherlands. Clin Nutr. 2003 Apr;22(2):147-52. doi: 10.1054/clnu.2002.0611. PMID 12706131
- [Background] Plank LD, Gane EJ, Peng S, Muthu C, Mathur S, Gillanders L, McIlroy K, Donaghy AJ, McCall JL. Nocturnal nutritional supplementation improves total body protein status of patients with liver cirrhosis: a randomized 12-month trial. Hepatology. 2008 Aug;48(2):557-66. doi: 10.1002/hep.22367. PMID 18627001